CLINICAL TRIAL: NCT05181007
Title: An Open-label, Two-stage Study Evaluating Drug-drug Interaction Between Ciprofol Injectable Emulsion and Mefanamic Acid or Valproate in Healthy Volunteers
Brief Title: Drug-drug Interaction Between Ciprofol and Mefanamic Acid or Valproate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HSK3486-111
Record Dates: First submitted 2021-12-01; First posted 2022-01-06 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Drug Drug Interaction
MeSH Terms: interventions — Mefenamic Acid; Valproic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MFA (Active Comparator): mefanamic acid
  Interventions: Drug: Mefanamic Acid
- VPA (Active Comparator): valproate
  Interventions: Drug: Valproate

INTERVENTIONS:
Drug: Mefanamic Acid — mefanamic acid once every 6 hours on Day 4 and Day 5, Ciprofol on Day 1 and Day 5
  Arms: MFA
Drug: Valproate — valproate once daily on Day 4 to Day 8, Ciprofol on Day 1 and Day 8
  Arms: VPA

SUMMARY:
study the effect of mefanamic acid or valproate on ciprofol

ELIGIBILITY:
Inclusion Criteria:

* Normal results of physical examination, laboratory tests (blood routine, blood biochemistry, and urine routine), and 12-lead ECG, or considered by the investigator to be clinically insignificant abnormalities; no significant potential difficult airway (modified Mallampati score Class I-II);
* No previous history of primary diseases in major organs, such as liver, kidneys, digestive tract, blood, and metabolic diseases; no history of malignant hyperthermia and other hereditary disorders; no history of mental/neurological disorders; no history of epilepsy; no contraindications for deep sedation/general anesthesia; no clinically significant history of anesthesia accidents;
* Understand procedures and methods of this trial, willing to sign the informed consent form and comply strictly with the clinical trial protocol to complete this study.

Exclusion Criteria:

* Known allergies to excipients of ciprofol injectable emulsion (soybean oil, glycerin, triglyceride, egg lecithin, sodium oleate, and sodium hydroxide), mefanamic acid, or valproate, or having contraindications to ciprofol/mefanamic acid/valproate; a history of drug allergies (including anesthetics), allergies, or prone to allergies;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
effect of mefanamic acid on the Cmax of ciprofol | 0-24hour post ciprofol dosing
  Peak Plasma Concentration (Cmax)
effect of mefanamic acid on the AUC of ciprofol | 0-24hour post ciprofol dosing
  Area under the plasma concentration versus time curve (AUC)
effect of valproate on the Cmax of ciprofol | 0-24hour post ciprofol dosing
  Peak Plasma Concentration (Cmax)
effect of valproate on the AUC of ciprofol | 0-24hour post ciprofol dosing
  Area under the plasma concentration versus time curve (AUC)

SECONDARY OUTCOMES:
Safety when ciprofol is co-administered with mefanamic acid or valproate | 0-24hour post ciprofol dosing
  Adverse event
effect of mefanamic acid or valproate on the MOAA/S of ciprofol | 0-24hour post ciprofol dosing
  MOAA/S
effect of mefanamic acid or valproate on the BIS of ciprofol | 0-24hour post ciprofol dosing
  BIS

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hospital Zhejiang University School of Medicine, Hanzhou, China